CLINICAL TRIAL: NCT02443389
Title: Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates
Acronym: AWAKEN
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); George Washington University (Other); McGill University (Other); Albert Einstein College of Medicine (Other); University of Rochester (Other); University of British Columbia (Other); University of Iowa (Other); University of Michigan (Other); University of New Mexico (Other); University of Virginia (Other); University of Washington (Other); University of Miami (Other); Case Western Reserve University (Other); University of Kentucky (Other); Maimonides Medical Center (Other); Stony Brook University (Other); The Canberra Hospital (Other); Children's Hospital Colorado (Other); St. Louis Children's Hospital (Other); Baylor College of Medicine (Other); Medanta, The Medicity, India (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, David Askenazi, MD, MsPH, Associate Professor, University of Alabama at Birmingham
Other Study IDs: X140917002
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury
Keywords: nephrotoxic; Fluid overload; Acute renal failure; Prematurity; Risk factors; Epidemiology
MeSH Terms: conditions — Acute Kidney Injury; Edema; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates admitted to NICU: Retrospective cohort of neonates admitted to NICU with stated inclusion and exclusion criteria

SUMMARY:
Introduction:

Based on single-center data, approximately 1 of every 3 newborns admitted to tertiary level neonatal intensive care units (NICU) develops acute kidney injury (AKI), and those with AKI have significantly worse outcomes. To stimulate discussion among researchers, the NIH NIDDK sponsored a workshop on neonatal AKI in April 2013. At that workshop, the group recognized the need to improve collaborations between neonatologists and nephrologists within and across centers. The investigators have created a multi-institutional, multi-disciplinary group, Neonatal Kidney Collaborative (NKC), in order to address the following critical needs identified at the workshop: AWAKEN is the inaugural study of this new collaboration.

1. Development of a standardized evidence-based definition of neonatal AKI
2. Evaluation of risk factors that predispose neonatal to AKI
3. Investigation into how fluid provision/ balance impacts biochemical and clinical outcomes

DETAILED DESCRIPTION:
The investigators will conduct a multi-center retrospective cohort study. The investigators will enroll eligible infants who meet inclusion and exclusion criteria at each center for 3 consecutive months. Based on average admissions for 2013 at our centers who meet inclusion and exclusion criteria, and estimate that it can enroll approximately 3000 infants during this time.

A. Specific Aim 1: Determine if the proposed neonatal AKI definition adapted to neonates is able to predict mortality, length of stay, and discharge serum creatinine (SCr).

1. Our primary hypothesis is that higher stages of AKI are associated with mortality, even after controlling for severity of illness, interventions and demographics.
2. Populations

   1. Inclusion Criteria - All infants born or admitted to a level 2 or 3 NICU will be screened. Infants who received intravenous fluids for > 48 hours will be eligible.
   2. Exclusion -- Infants admitted to the NICU at 2 weeks of age or older; Infants who undergo cardiovascular surgery repair of a congenital heart lesion within 1 week of life; Infants diagnosed with a lethal anomaly upon admission; Infants who die within 48 hours after birth
3. Primary Exposure - Neonatal AKI definitions (table 3)
4. Primary Outcome - Survival

   1. In premature infants - defined as survival to 36 weeks post gestational age or hospital discharge (whichever comes first)
   2. In term infants - defined as hospital survival to 28 days.
5. Secondary outcomes

   1. Hospital length of stay
   2. Last serum creatinine obtained
6. Potential confounders - gestational age, birth weight, 5 minute APGAR score, multiple gestation, significant renal anomalies, SNAP-II score
7. Exploratory outcomes - recognize that the proposed definition may not be the best definition to predict clinical outcomes. Also recognize that there may be a need to have different definitions for premature infants. The investigators plan to explore how other definitions reported in the literature can predict these outcomes (for example using the 90th % for normative values). In addition, this will have the largest comprehensive database to explore new definitions which could incorporate urine output, fluid balance and other factors.

B. Specific Aim 2: Define the risk factors associated with neonatal AKI.

1. Our hypothesis is that maternal and infant risk factors will predict AKI.
2. Population - same as in Specific Aim 1
3. Design - randomize cohort to a prediction and a validation groups. Develop a risk factor prediction model with the first group, and test the ability of the model to predict AKI with the second group.
4. Exposures (see full list in appendix 1 - Data collection sheets)

   1. Maternal Demographic Factors
   2. Neonatal Demographic Factors
   3. Interventions / Medications
   4. Co-Morbidities
5. Primary Outcome - KDIGO AKI definition modified for neonates (Table 3).

C. Specific Aim 3: Determine how fluid balance during the first few weeks of life relates to biochemical data and clinical outcomes.

1. Our hypotheses are that fluid provision affects chemistry panels (serum creatinine, blood urea nitrogen, serum sodium) and that fluid balance is associated with clinical outcomes.
2. Population - same as in Specific Aim 1
3. Design

   1. Evaluation of fluid balance - will use birth weight as the reference weight and calculate changes in weight over time as a percentage of birth weight.
   2. Will describe the association between fluid balance and changes in serum creatinine (SCr), blood urea nitrogen (BUN) and serum sodium.
   3. Will then evaluate how fluid balance (and the associated biochemical changes) affects clinical outcomes.
4. Primary Clinical Outcome - Survival

   1. In premature infants - defined as survival to 36 weeks post gestational age or hospital discharge (whichever comes first)
   2. In term infants - defined as hospital survival to 28 days.
5. Secondary outcomes

   1. Hospital length of stay
   2. Ventilator free days in the first 28 days of life.
   3. Bronchopulmonary dysplasia
   4. Intraventricular hemorrhage
   5. Last serum creatinine obtained
   6. Use of blood pressure support medications
   7. Use of diuretics
   8. Patent ductus arteriosus

Data will be captured at each institution and entered into web-based forms in real time.

The investigators plan to have 5 different integrated forms:

1. Screening form
2. Baseline form for included infants
3. Daily Assessment form (first 7 days after birth)
4. Weekly Assessment form (weeks 2 - 18)
5. Discharge form

ELIGIBILITY:
Inclusion Criteria:

1. All infants born or admitted to a level 2 or 3 NICU will be screened.
2. Infants who received intravenous fluids for > 48 hours will be eligible.

Exclusion Criteria:

1. Infants admitted to the NICU at 2 weeks of age or older
2. Infants who undergo cardiovascular surgery repair of a congenital heart lesion within 1 week of life
3. Infants diagnosed with a lethal anomaly upon admission
4. Infants who die within 48 hours after birth

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will conduct a multi-center retrospective cohort study. The investigators will enroll eligible infants who meet inclusion and exclusion criteria at each center for 3 consecutive months. Based on average admissions for 2013 at our centers who meet inclusion and exclusion criteria, it is estimated that it can enroll approximately 3000 infants during this time. All infants admitted to the NICU between January 1, 2014 and march 31, 2014 will be screened for the study.
Sampling Method: Non-Probability Sample
Enrollment: 2186 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Determine if the KDIGO AKI definition adapted to neonates can predict mortality, length of stay, and discharge serum creatinine (SCr). | NICU admit though 18 weeks hospitalization or hospital discharge whichever comes first.
Define the major risk factors associated with neonatal AKI. We will randomly split the cohort into two groups. We will develop a risk factor prediction model with the first group, and test the ability of the model to predict AKI with the second group. | NICU admit though 18 weeks hospitalization or hospital discharge whichever comes first.
Determine how fluid balance during the first few weeks of life relates to biochemical data and clinical outcomes. | NICU admit though 18 weeks hospitalization or hospital discharge whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: David Askenazi, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selewski DT, Gist KM, Nathan AT, Goldstein SL, Boohaker LJ, Akcan-Arikan A, Bonachea EM, Hanna M, Joseph C, Mahan JD, Mammen C, Nada A, Reidy K, Staples A, Wintermark P, Griffin R, Askenazi DJ, Guillet R; Neonatal Kidney Collaborative. The impact of fluid balance on outcomes in premature neonates: a report from the AWAKEN study group. Pediatr Res. 2020 Feb;87(3):550-557. doi: 10.1038/s41390-019-0579-1. Epub 2019 Sep 19. PMID 31537009
- [Background] Starr MC, Boohaker L, Eldredge LC, Menon S, Griffin R, Mayock D, Askenazi D, Hingorani S; Neonatal Kidney Collaborative. Acute Kidney Injury is Associated with Poor Lung Outcomes in Infants Born >/=32 Weeks of Gestational Age. Am J Perinatol. 2020 Jan;37(2):231-240. doi: 10.1055/s-0039-1698836. Epub 2019 Nov 18. PMID 31739364
- [Background] Askenazi D, Abitbol C, Boohaker L, Griffin R, Raina R, Dower J, Davis TK, Ray PE, Perazzo S, DeFreitas M, Milner L, Ambalavanan N, Cole FS, Rademacher E, Zappitelli M, Mhanna M; Neonatal Kidney Collaborative. Optimizing the AKI definition during first postnatal week using Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates (AWAKEN) cohort. Pediatr Res. 2019 Feb;85(3):329-338. doi: 10.1038/s41390-018-0249-8. Epub 2018 Dec 13. PMID 30643188
- [Background] Charlton JR, Boohaker L, Askenazi D, Brophy PD, D'Angio C, Fuloria M, Gien J, Griffin R, Hingorani S, Ingraham S, Mian A, Ohls RK, Rastogi S, Rhee CJ, Revenis M, Sarkar S, Smith A, Starr M, Kent AL; Neonatal Kidney Collaborative. Incidence and Risk Factors of Early Onset Neonatal AKI. Clin J Am Soc Nephrol. 2019 Feb 7;14(2):184-195. doi: 10.2215/CJN.03670318. Epub 2019 Jan 31. PMID 31738181
- [Background] Harer MW, Askenazi DJ, Boohaker LJ, Carmody JB, Griffin RL, Guillet R, Selewski DT, Swanson JR, Charlton JR; Neonatal Kidney Collaborative (NKC). Association Between Early Caffeine Citrate Administration and Risk of Acute Kidney Injury in Preterm Neonates: Results From the AWAKEN Study. JAMA Pediatr. 2018 Jun 4;172(6):e180322. doi: 10.1001/jamapediatrics.2018.0322. Epub 2018 Jun 4. PMID 29610830
- [Background] Kraut EJ, Boohaker LJ, Askenazi DJ, Fletcher J, Kent AL; Neonatal Kidney Collaborative (NKC). Incidence of neonatal hypertension from a large multicenter study [Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates-AWAKEN]. Pediatr Res. 2018 Aug;84(2):279-289. doi: 10.1038/s41390-018-0018-8. Epub 2018 May 23. PMID 29795211
- [Background] Jetton JG, Boohaker LJ, Sethi SK, Wazir S, Rohatgi S, Soranno DE, Chishti AS, Woroniecki R, Mammen C, Swanson JR, Sridhar S, Wong CS, Kupferman JC, Griffin RL, Askenazi DJ; Neonatal Kidney Collaborative (NKC). Incidence and outcomes of neonatal acute kidney injury (AWAKEN): a multicentre, multinational, observational cohort study. Lancet Child Adolesc Health. 2017 Nov;1(3):184-194. doi: 10.1016/S2352-4642(17)30069-X. PMID 29732396
- [Background] Selewski DT, Akcan-Arikan A, Bonachea EM, Gist KM, Goldstein SL, Hanna M, Joseph C, Mahan JD, Nada A, Nathan AT, Reidy K, Staples A, Wintermark P, Boohaker LJ, Griffin R, Askenazi DJ, Guillet R; Neonatal Kidney Collaborative. The impact of fluid balance on outcomes in critically ill near-term/term neonates: a report from the AWAKEN study group. Pediatr Res. 2019 Jan;85(1):79-85. doi: 10.1038/s41390-018-0183-9. Epub 2018 Sep 20. PMID 30237572
- [Background] Kirkley MJ, Boohaker L, Griffin R, Soranno DE, Gien J, Askenazi D, Gist KM; Neonatal Kidney Collaborative (NKC). Acute kidney injury in neonatal encephalopathy: an evaluation of the AWAKEN database. Pediatr Nephrol. 2019 Jan;34(1):169-176. doi: 10.1007/s00467-018-4068-2. Epub 2018 Aug 28. PMID 30155763
- [Background] Charlton JR, Boohaker L, Askenazi D, Brophy PD, Fuloria M, Gien J, Griffin R, Hingorani S, Ingraham S, Mian A, Ohls RK, Rastogi S, Rhee CJ, Revenis M, Sarkar S, Starr M, Kent AL; Neonatal Kidney Collaborative (NKC). Late onset neonatal acute kidney injury: results from the AWAKEN Study. Pediatr Res. 2019 Feb;85(3):339-348. doi: 10.1038/s41390-018-0255-x. Epub 2018 Dec 13. PMID 30546043
- [Background] Jetton JG, Guillet R, Askenazi DJ, Dill L, Jacobs J, Kent AL, Selewski DT, Abitbol CL, Kaskel FJ, Mhanna MJ, Ambalavanan N, Charlton JR; Neonatal Kidney Collaborative. Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates: Design of a Retrospective Cohort Study. Front Pediatr. 2016 Jul 19;4:68. doi: 10.3389/fped.2016.00068. eCollection 2016. PMID 27486571
- [Background] Kent AL, Charlton JR, Guillet R, Gist KM, Hanna M, El Samra A, Fletcher J, Selewski DT, Mammen C. Neonatal Acute Kidney Injury: A Survey of Neonatologists' and Nephrologists' Perceptions and Practice Management. Am J Perinatol. 2018 Jan;35(1):1-9. doi: 10.1055/s-0037-1604260. Epub 2017 Jul 14. PMID 28709164
- [Background] Stoops C, Boohaker L, Sims B, Griffin R, Selewski DT, Askenazi D; on behalf of the National Kidney Collaborative (NKC). The Association of Intraventricular Hemorrhage and Acute Kidney Injury in Premature Infants from the Assessment of the Worldwide Acute Kidney Injury Epidemiology in Neonates (AWAKEN) Study. Neonatology. 2019;116(4):321-330. doi: 10.1159/000501708. Epub 2019 Aug 28. PMID 31461717